CLINICAL TRIAL: NCT06166680
Title: Assessment of Tongue Motor Functions in Healthy Children
Brief Title: Tongue Muscular Assessment in Healthy Children
Acronym: TMAC
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, Prof., Université Catholique de Louvain
Other Study IDs: TMAC
Record Dates: First submitted 2023-11-22; First posted 2023-12-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Tongue; Motor functions
MeSH Terms: interventions — Anthropometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy children: Healthy children between the ages of 4 to 17 will undergo tongue motor functions assessment and their parents will fulfill the Pediatric Sleep Questionnaire
  Interventions: Other: Sleep quality assessment; Other: Anthropometry; Other: Tongue strength assessment; Other: Tongue endurance assessment; Other: Orofacial praxis assessment

INTERVENTIONS:
Other: Sleep quality assessment — The following item will be assessed in all subjects (n=420):
  1. Sleep, through the Pediatric Sleep Questionnaire.
Other: Anthropometry — The following items will be assessed in all subjects (n=420):
  2. Anthropometric data : 2.1 Height; 2.2 Weight; 2.3 Maximal mouth opening; 2.4 Maximal mouth opening with tongue to palate (with the Quick Tongue-Tie assessment tool)
Other: Tongue strength assessment — The following items will be assessed in all subjects (n=420):
  3. Tongue pressure (in kPa) exerted against the IOPI (Iowa Oral Performance Instrument) bulb while swallowing.
  4. Tongue peak pressure (i.e., the maximal pressure - Pmax - exerted against the IOPI bulb) during 3 sec. of tongue elevation.
  5. Tongue peak pressure during 3 sec. of tongue protrusion.
Other: Tongue endurance assessment — The following items will be assessed in all subjects (n=420):
  6. The tongue endurance (i.e., the time to task failure in maintaining a pressure equal to 50%Pmax against the IOPI bulb) during tongue elevation.
  7. The tongue endurance during tongue protrusion.
Other: Orofacial praxis assessment — - The following item will be assessed in a subset of subjects (n=31): 8. Orofacial praxis through the Motricité Bucco-Linguo-Faciale (MBLF) test.

SUMMARY:
This study aims to obtain normative values for tongue motor functions in healthy children.

DETAILED DESCRIPTION:
Since the tongue is a complex structure consisting of a continuous array of muscle fibers with varying orientation, tongue motor functions (strength, endurance) are likely to differ according to a protrusion (pulling out the tongue), elevation (lifting the tongue to the roof of the mouth) or swallowing movement.

There are currently no normative data for the motor functions of the tongue in children. After their parents fulfilled the Pediatric Sleep Questionnaire, each included children will undergo an anthropometric and a tongue motor functions assessment.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 4 and 17

Exclusion Criteria:

* Eating disorder
* Dysphagia
* Cardiorespiratory disorder
* Neurological disorder (including neuromuscular disorders)
* Previous or ongoing obstructive sleep apnea-hypopnea syndrome
* Previous or ongoing cancer of the head or neck
* Previous oral or pharyngeal surgery (except for the surgical removal of wisdom teeth)
* Cranial, oral or upper airway malformation (ex.: nasal cavities, pharynx)
* Previous or ongoing orthodontic treatment (e.g. braces)
* More than 33% of positive answers to the Pediatric Sleep Questionnaire (8/22)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children between the ages of 4 to 17
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Tongue peak pressure during elevation and protrusion movements | At baseline
  Tongue peak pressure during elevation and protrusion movements will be measured via the IOPI (Iowa Oral Performance Instrument) device

SECONDARY OUTCOMES:
Tongue mobility restriction | At baseline
  Assessed through the ratio between maximal mouth opening and maximal mouth opening with tongue to palate, measured with the Quick Tongue-Tie Assessment tool
Orofacial praxis | At baseline
  In a subset of subjects (n=31), orofacial praxis will be assessed through the Motricité Bucco-Linguo-Faciale (MBLF) test
Tongue endurance during elevation and protrusion movements | At baseline
  Tongue endurance during elevation and protrusion movements will be measured via the IOPI device and a timer
Tongue pressure during swallowing | At baseline
  Tongue pressure during swallowing will be measured via the IOPI device

CONTACTS AND LOCATIONS:
Overall Officials: William Poncin, PT, PhD, Prof, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Woluwe-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: No